CLINICAL TRIAL: NCT06679322
Title: A Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase IIb Clinical Trial of Androtriol Injection for the Treatment of Acute Ischemic Stroke
Brief Title: The Androtriol Injection for the Treatment of Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YC-6-PIIb-AIS
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Androtriol; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (high-dose group) (Experimental): Androtriol injection (300 mg BID)
  Interventions: Drug: Androtriol Injection (High-dose group)
- Intervention Group (low-dose group) (Experimental): Androtriol injection (100 mg BID)
  Interventions: Drug: Androtriol Injection (Low-dose group)
- Placebo (Placebo Comparator): Hydroxypropyl-β-cyclodextrin injection
  Interventions: Drug: Hydroxypropyl-β-cyclodextrin injection

INTERVENTIONS:
Drug: Androtriol Injection (High-dose group) — Participants will receive 30 mL of Androtriol Injection per dose, administered every 12 hours for 7 consecutive days. Each infusion will be administered over a period of 30±5 minutes.
  Arms: Intervention Group (high-dose group)
Drug: Androtriol Injection (Low-dose group) — Participants will receive 10 mL of Androtriol Injection combined with 20 mL of placebo (Hydroxypropyl Beta-Cyclodextrin Injection) per dose, administered every 12 hours for 7 consecutive days. Each infusion will be administered over a period of 30±5 minutes.
  Arms: Intervention Group (low-dose group)
Drug: Hydroxypropyl-β-cyclodextrin injection — Participants will receive 30 mL of Hydroxypropyl-β-cyclodextrin injection per dose, administered every 12 hours for 7 consecutive days. Each infusion will be completed within 30±5 minutes.
  Arms: Placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, phase IIb clinical trial of Androtriol injection for the treatment of acute ischemic stroke. The goal of this trial is to explore the efficacy and safety of different doses of Androtriol injection in patients with acute ischemic stroke (AIS) who received vascular recanalization treatment within 24 hours of symptom onset.

Participants will receive a low-dose Androtriol injection (100 mg BID), a high-dose Androtriol injection (300 mg BID), or a placebo intravenously within 24 hours of stroke onset. They will be treated twice daily (every 12 hours) for 7 days, with a total of 14 doses over the course of the study. Each infusion will last approximately 30±5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 80 years, male or female；
2. mRS score ≤1 prior to this onset;
3. Planning to receive or have received intravascular recanalization therapy at our center within 24h of onset;
4. To complete the first administration of the investigational medication within 24h of onset;
5. NIHSS（National Institutes of Health Stroke Scale）score≥6 prior to intravascular recanalization;
6. Informed consent.

Exclusion Criteria:

1. Intracranial hemorrhagic diseases, including hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.;
2. Severe disorders of consciousness: NIHSS 1a≥2 points;
3. Large infarct core (ASPECTS <6, or>1/3 of MCA territory involved, as evidenced by CT or MRI);
4. Severe hypertension: systolic blood pressure ≥185mmHg or diastolic blood pressure ≥110mmHg after medication control;
5. History of severe kidney disease (such as dialysis), or eGFR <45 mL/min/1.73m²;
6. History of severe liver disease, or ALT, AST levels more than 3 times of the upper limit of normal, or bilirubin more than 3 times of the upper limit of normal;
7. Cardiovascular diseases, such as complete atrioventricular block, history of congestive heart failure (CHF), or heart function classification≥NYHA Class III;
8. Critically ill patients with an expected lifespan≤90 days;
9. History of epilepsy or epilepsy-like symptoms during stroke or severe psychiatric disorders, intellectual disability, or dementia;
10. History of intracranial hemorrhage;
11. Severe injury or surgery history within 3 months of onset;
12. Have received>1 dose of neuroprotective drugs after this onset, such as edaravone, edaravone dexborneol injection, ginkgo lactone, ginkgo diterpene glucamine，etc;
13. Allergy to the investigational drug (either the active ingredient androtriol or the excipient hydroxypropyl beta-cyclodextrin) or similar chemical structure drugs;
14. Pregnant or breastfeeding;
15. Participation in other clinical trials within 3 months of onset;
16. Unsuitable for participating in this study judged by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with a modified Rankin Scale (mRS) score of 0-1 at 90 days after stroke onset | 90 days after stroke onset
  The mRS denotes modified Rankin Scale, ranging from 0 (no neurologic deficit, no symptoms or completely recovered) to 6 (death).

SECONDARY OUTCOMES:
The modified Rankin Scale (mRS) scores at 90 days after stroke | 90 days after stroke onset
  The mRS denotes modified Rankin Scale, ranging from 0 (no neurologic deficit, no symptoms or completely recovered) to 6 (death).
The proportion of participants with a modified Rankin Scale (mRS) score of 0-2 at 90 days after stroke onset | 90 days after stroke onset
  The mRS denotes modified Rankin Scale, ranging from 0 (no neurologic deficit, no symptoms or completely recovered) to 6 (death).
The change of the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 14 days after stroke onset or at discharge | Baseline, 14 days or at discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe stroke.
The change of Barthel Index (BI) scores at 30 days and 90 days after stroke onset | Baseline, 30 days and 90 days after stroke onset
  The Barthel Index for Activities of Daily Living (ADL) assesses functional independence, generally in stroke patients. The higher the score, the more independent the patient is in completing the measured ADLs.
The change of EuroQol Five Dimensions Questionnaire (EQ-5D) scores at 30 days and 90 days after stroke onset | Baseline, 30 days and 90 days after stroke onset
  The EQ-5D assesses quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is scored on a scale from 1 to 3, with lower scores (closer to 1) indicating better health outcomes.

OTHER OUTCOMES:
Incidence of adverse events (AE) and treatment-related adverse events (TEAE) | From the time of administration to day 90
Incidence of significant adverse events and serious adverse events (SAE) | From the time of administration to day 90
Symptomatic intracranial hemorrhage (sICH) within 36 hours after thrombolysis (SITS-MOST criteria) | 36 hours after thrombolysis
  The Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) criteria: Within 36 hours after thrombolysis, an increase of NIHSS score≥4 compare to baseline or the lowest NIHSS, with > 30% infarction area.
All-cause mortality | From the time of administration to day 90
Discontinuation of medication due to any reason or adverse events | From the time of administration to day 90
The change of midline shift from baseline at 22-36 hours and 7 days after first treatment | Baseline, 22-36 hours, and 7 days after first treatment
The change of lesion volume from baseline at 22-36 hours and 7 days after first treatment | Baseline, 22-36 hours, and 7 days after first treatment
The change of edema volume on the lesion side from baseline at 22-36 hours and 7 days after first treatment | Baseline, 22-36 hours, and 7 days after first treatment

IPD SHARING:
Plan to Share IPD: No